CLINICAL TRIAL: NCT04319159
Title: An Open-label Phase I Study to Evaluate the Pharmacokinetics of 5-aminolevulinic Acid and Protoporphyrin IX in Human Plasma Under Maximal Use Conditions After Topical Application of 3 Tubes of BF-200 ALA 10% Gel for Photodynamic Therapy (PDT) in Subjects Suffering From Actinic Keratosis
Brief Title: Study to Evaluate the Safety of BF-200 ALA (Ameluz®) for Photodynamic Therapy (PDT) in the Treatment of Expanded Fields of Actinic Keratosis (AK)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biofrontera Bioscience GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALA-AK-CT015
Record Dates: First submitted 2020-03-10; First posted 2020-03-24 (Actual); Results first posted 2021-11-11 (Actual); Last update posted 2021-11-11 (Actual); Status verified 2021-10

CONDITIONS: Actinic Keratoses
Keywords: Actinic keratosis; Photodynamic therapy; 5-aminolevulinic acid; Protoporphyrin IX; Pharmacokinetics
MeSH Terms: conditions — Keratosis, Actinic | interventions — BF-200 ALA

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- BF-200 ALA (Experimental): Topical application of BF-200 ALA containing 7.8% 5-ALA (5-aminolevulinic acid).
  One single Photodynamic therapy (PDT).
  Interventions: Combination Product: BF-200 ALA and red light LED lamp

INTERVENTIONS:
Combination Product: BF-200 ALA and red light LED lamp — Combination Product: Photodynamic therapy (PDT) using BF-RhodoLED® (ALA-PDT, Ameluz®-PDT).

SUMMARY:
The aim of this study is to assess the pharmacokinetics (PK) of the parent drug 5-aminolevulinic acid (ALA) and its active metabolite protoporphyrin IX (PpIX) during photodynamic therapy with 3 tubes of BF-200 ALA 10% gel (Ameluz®) in combination with the BF-RhodoLED® lamp in the systemic circulation of diseased individuals presenting with actinic keratosis (AK) on the face/scalp or in the periphery (neck/trunk/extremities) along with subjects' safety/tolerability during and after treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with at least 12 distinctive and clinically confirmed mild to severe AK lesions (according to Olsen et al. 1991 (37)) with a diameter of ≥ 4 mm each, on either the face/scalp (including forehead, excluding eyes, nostrils, ears, and mouth) or the neck/trunk/extremities, within treatment field(s) of about 60 cm² in total. Treatment field(s) may be discontinuous but must be within 2 illumination areas of the BF-RhodoLED® lamp (6 cm x 16 cm each).
2. All genders 18-85 years of age (inclusive).
3. Willingness and ability of the subject to provide informed consent and to sign the Health Insurance Portability and Accountability Act (HIPAA) form. A study-specific informed consent form and HIPAA form must be obtained in writing for all subjects prior to starting any study procedures.
4. Willingness and ability to comply with study procedures, particularly willingness to receive one PDT with up to two illumination devices simultaneously.
5. Subjects with good general health and subjects with clinically stable medical conditions will be permitted to be included in the study.
6. Subjects receiving any drugs affecting coagulation (e.g. anticoagulants, anti-platelet drugs) should be on a stable dose.
7. Acceptance to abstain from extensive sunbathing and the use of solarium during the clinical study.
8. Women of child-bearing potential must have a negative serum pregnancy test and must use an adequate and highly effective or two effective methods of contraception throughout the study.

Exclusion Criteria:

1. Any known history of hypersensitivity to ALA, porphyrins or excipients of BF- 200 ALA.
2. History of soy or peanut allergy.
3. Subjects with sunburn within illumination areas (reassessment of subjects is allowed once if the sunburn is expected to resolve within the screening period. Reassessment can be done on the day of the actual treatment.).
4. Clinically significant medical conditions making implementation of the protocol or interpretation of the study results difficult or impairing subjects' safety such as:

   1. Presence of porphyria or known photodermatoses
   2. Known diagnosis of human immunodeficiency virus (HIV) based on clinical history
   3. Metastatic tumor or tumor with high probability of metastasis
   4. Infiltrating skin neoplasia (suspected or known)
   5. Unstable cardiovascular disease (New York Heart Association [NYHA] class III, IV)
   6. Unstable hematologic (including Myelodysplastic syndrome), hepatic, renal, neurologic, or endocrine condition
   7. Unstable collagen-vascular condition
   8. Unstable gastrointestinal condition
   9. Immunosuppressive condition
   10. Presence of clinically significant inherited or acquired coagulation defect
5. Clinical diagnosis of atopic dermatitis, Bowen's disease, BCC, eczema, psoriasis, rosacea, SCC, other malignant or benign tumors in the treatment field(s), or other possible confounding skin conditions (e.g. wounds, irritations, bleeding or skin infections) within or in close proximity (< 5 cm distance) to treatment field(s). (Reassessment of subjects is allowed once if wounds, irritations, bleeding or skin infections are expected to resolve within the screening period. Reassessment can be done on the day of the actual treatment.)
6. Presence of strong pigmentation, tattoos or any other abnormality that may impact lesion assessment or light penetration in the treatment field(s).
7. More than moderate smoker (e.g. > 10 cigarettes/day or equivalent).
8. Suspicion of drug or alcohol abuse. For the purpose of this study, alcohol abuse is defined as more than moderate alcohol consumption (> 1 drink/day for women and > 2 drinks/day for men).
9. Physical treatment of malignant or benign tumors of the skin within the treatment field(s) and at a distance of < 5 cm to the treatment field(s) during the last 4 weeks prior to screening.
10. Any therapy such as cryotherapy, laser therapy, electrodessication, surgical removal of lesions, curettage, or treatment with chemical peels such as trichloroacetic acid within the treatment field(s), or within a radius less than 5 cm away from the treatment field(s) 4 weeks prior to screening.
11. Any topical medical treatment of the skin within the designated time period below:

    1. Topical treatment with ALA or methyl-aminolevulinate (MAL) or an investigational drug in- and outside the treatment field(s) within 8 weeks prior to screening.
    2. Topical treatment with immunomodulatory/immunosuppressive antiinflammatory, or cytotoxic agents inside the treatment field(s) or within a radius less than 5 cm away from the treatment field(s) within 8 weeks prior to screening.
    3. Start of topical administration of medication with hypericin or other drugs with phototoxic or photoallergic potential in- and outside the treatment field(s) within 8 weeks prior to screening. Subjects may, however, be eligible if such medication was applied for more than 8 weeks prior to screening visit without evidence of an actual phototoxic/photoallergic reaction.
12. Any use of the below specified systemic treatments within the designated periods:

    1. Use of cytotoxic drugs within 24 weeks, immunomodulators or immunosuppressive therapies or use of ALA or ALA-esters (e.g. MAL) within 12 weeks, investigational drugs or drugs known to have major organ toxicity within 8 weeks, interferon or corticosteroids (oral or injectable) within 6 weeks prior to screening.
    2. Start of intake of medication with hypericin or systemically-acting drugs with phototoxic or photoallergic potential within 8 weeks prior to screening. Subjects may, however, be eligible if such medication was taken in or applied for more than 8 weeks prior to screening visit without evidence of an actual phototoxic/photoallergic reaction.
13. Laboratory values outside the reference range that are clinically significant in the opinion of the investigator (e.g., suggesting an unknown disease and requiring further clinical evaluation according to investigator), especially aspartate aminotransferase (AST), alanine aminotransferase (ALT), gamma glutamyl transpeptidase (gamma- GT).
14. Impaired renal function (Glomerular filtration rate below 50 mL/min/1.73m² estimated by Modification of Diet in Renal Disease equation (MDRD)).
15. Positive test for HIV antibodies, Hepatitis B-virus surface antigen (HBsAg) or positive Anti-hepatitis C-virus antibody (Anti-HCV) test.
16. Significant blood donation or blood loss (≥ 500 mL) within three months prior to Visit 2.
17. Breast-feeding women.
18. Subject unlikely to comply with the protocol, e.g. inability to return for visits, unlikely to complete the study, or inappropriate in the opinion of the investigator.
19. Prior participation in the study (participation is defined as having been screened).
20. A member of study site staff or sponsor staff directly involved in the conduct of the protocol or a close relative thereof.
21. Simultaneous participation in a further clinical study.

Reassessment of subjects is allowed once if sunburn, wounds, irritations, bleeding or skin infections detected at Visit 1 are expected to resolve within the screening period.

Reassessment can be done on the day of the actual treatment.

Dosing day exclusion criteria:

1. Febrile or infectious illness within 7 days prior to Visit 2.
2. Subjects with sunburn, wounds, irritations, bleeding or other confounding skin conditions within illumination areas at Visit 2.
3. Use of topical NSAIDs inside and outside the treatment field(s) or systemic intake of NSAIDs within 7 days prior to Visit 2.

In case a subject meets one of the dosing day exclusion criteria, Visit 2 can be rescheduled once within 14 days. Meeting any of the dosing day exclusion criteria on the rescheduled visit will lead to discontinuation of the trial.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2020-03-05 (Actual); Primary Completion 2020-09-09 (Actual); Study Completion 2020-10-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- DermResearch Inc., Austin, Texas, United States

REFERENCES:
- [Derived] Novak B, DuBois J, Chahrour O, Papusha T, Hirt S, Philippi T, Zogel C, Osenberg K, Schmitz B, Lubbert H. Clinical Pharmacokinetics and Safety of a 10% Aminolevulinic Acid Hydrochloride Nanoemulsion Gel (BF-200 ALA) in Photodynamic Therapy of Patients Extensively Affected With Actinic Keratosis: Results of 2 Maximal Usage Pharmacokinetic Trials. Clin Pharmacol Drug Dev. 2022 Apr;11(4):535-550. doi: 10.1002/cpdd.1023. Epub 2021 Oct 11. PMID 34633154

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Trial was conducted at one site in the USA that recruited subjects. Recruitment of subjects started on 05 March 2020.
Pre-assignment Details: 48 subjects were screened for eligibility which was within 2 weeks prior to PDT. 2 of 48 subjects were re-screened due to the COVID-19 implications. 13 subjects were excluded as screening failures and one subject withdrew informed consent before treatment. In total, 32 subjects were treated. In this single-arm study, all participants received identical active treatment. Study data were analyzed primarily overall and additionally according to strata.
Groups:
- BF-200 ALA (Stratum Face/Scalp and Stratum Periphery): • Topical application of BF-200 ALA containing 7.8% 5-ALA (5-aminolevulinic acid) • Each subject received three entire tubes of the IMP (2 g each, containing 156 mg ALA), resulting in a total dose of 468 mg ALA (free base) • The amount was sufficient to cover one treatment field (continuous field or discontinuous field with several patches), totaling approx. 60 cm² with BF-200 ALA gel at a thickness of approx. 1 mm • Treatment field(s) could be located on either the face/scalp or in the periphery (neck/trunk/extremities) excluding the genitalia (minimal distance of about 1 cm) • IMP dried for approx. 10 min • Subjects had to stay in a well-tempered environment during 3h incubation under light-blocking, occlusive dressing • Dressing was removed; remnant gel wiped off • Illumination with BF-RhodoLED® (10 min; 37 J/cm²) • In case of discontinuous treatment field(s), two BF-RhodoLED® lamps were used simultaneously • One single PDT was performed
Period: Overall Study
Arm/Group | BF-200 ALA (Stratum Face/Scalp and Stratum Periphery)
Started | 48
Completed | 32
Not Completed | 16
Not completed — Screening failure | 13
Not completed — Re-screening due to COVID-19 implications | 2
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- Stratum: Face/Scalp; Stratum: Periphery: • Topical application of BF-200 ALA containing 7.8% 5-ALA (5-aminolevulinic acid) • Each subject received three entire tubes of the IMP (2 g each, containing 156 mg ALA), resulting in a total dose of 468 mg ALA (free base) • The amount was sufficient to cover one treatment field (continuous field or discontinuous field with several patches), totaling approx. 60 cm² with BF-200 ALA gel at a thickness of approx. 1 mm • Treatment field(s) could be located on either the face/scalp or in the periphery (neck/trunk/extremities) excluding the genitalia (minimal distance of about 1 cm) • IMP dried for approx. 10 min • Subjects had to stay in a well-tempered environment during 3h incubation under light-blocking, occlusive dressing • Dressing was removed; remnant gel wiped off • Illumination with BF-RhodoLED® (10 min; 37 J/cm²) • In case of discontinuous treatment field(s), two BF-RhodoLED® lamps were used simultaneously • One single PDT was performed
- Total: Total of all reporting groups
Arm/Group | Stratum: Face/Scalp | Stratum: Periphery | Total
Number analyzed (Participants) | 16 | 16 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.8 (6.0) | 63.8 (6.1) | 64.3 (6.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 6 | 7
  Male | 15 | 10 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 15 | 15 | 30
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 16 | 16 | 32
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 16 | 16 | 32
Fitzpatrick skin type [Count of Participants; unit: Participants] — Subjects' skin type was assessed at the screening visit using a six-level Fitzpatrick Skin Type Rating Scale, which ranges from very fair (skin type I) to very dark (skin type VI).
  Participants
    I | 6 | 13 | 19
    II | 8 | 3 | 11
    III | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Assessment of Baseline-adjusted Plasma Concentration-time Curves for ALA After a Single PDT Treatment Applying 3 Tubes of BF-200 ALA in Conjunction With the BF-RhodoLED® Under Maximal Use Conditions in Subjects With Mild to Severe Actinic Keratosis.
Description: Blood samples for ALA analysis for each subject were collected, starting at Visit 1 and then 0.5h prior to BF-200 ALA application for up to 10h afterwards. The concentrations of ALA in plasma were measured by an analytical laboratory using validated, internally standardized liquid chromatography-tandem mass spectrometry methods.
Time Frame: On treatment day (day 0): 0.5, 1, 1.5, 2, 2.5, 3*, 3.5, 4, 5, 6, 8, 10 hours post-dose (*prior to illumination)
Population: ALA Pharmacokinetic Set (PKS ALA): includes all subjects who had at least one evaluable pre-dose and post-dose pharmacokinetic sample (i.e., samples taken after the application of BF-200 ALA); a pre-dose/post-dose sample was regarded evaluable if the plasma concentration was at or above LLOQ.
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | Stratum: Face/Scalp | Stratum: Periphery
Number analyzed (Participants) | 16 | 16
ng/mL
  0.5h | 8.904 (3.3502) | 10.21 (5.2811)
  1h | 12.45 (3.1865) | 9.383 (5.2972)
  1.5h | 18.96 (2.4231) | 10.15 (4.3289)
  2h | 18.02 (2.7917) | 9.561 (6.3130)
  2.5h | 23.06 (2.1768) | 6.233 (5.7572)
  3h | 24.71 (2.2076) | 13.55 (5.3204)
  3.5h | 22.00 (1.9477) | 10.77 (3.3921)
  4h | 16.54 (1.7954) | 7.172 (3.4656)
  5h | 10.21 (1.6002) | 4.558 (2.1024)
  6h | 5.812 (2.2470) | 4.231 (1.9599)
  8h | 3.250 (2.0091) | 2.871 (1.9438)
  10h | 2.536 (2.0871) | 3.444 (1.8003)

2. Primary Outcome: Assessment of Baseline-adjusted Plasma Concentration-time Curves for PpIX After a Single PDT Treatment Applying 3 Tubes of BF-200 ALA in Conjunction With the BF-RhodoLED® Under Maximal Use Conditions in Subjects With Mild to Severe Actinic Keratosis.
Description: Blood samples for PpIX analysis for each subject were collected, starting at Visit 1 and then 0.5h prior to BF-200 ALA application for up to 10h afterwards. The concentrations of PpIX in plasma were measured by an analytical laboratory using validated, internally standardized liquid chromatography-tandem mass spectrometry methods.
Time Frame: On treatment day (day 0): 0.5, 1, 1.5, 2, 2.5, 3*, 3.5, 4, 5, 6, 8, 10 hours post-dose (*prior to illumination)
Population: PpIX Pharmacokinetic Set (PKS PpIX): includes all subjects who had at least one evaluable pre-dose and post-dose pharmacokinetic sample (i.e., samples taken after the application of BF-200 ALA); a pre-dose/post-dose sample was regarded evaluable if the plasma concentration was at or above LLOQ.
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | Stratum: Face/Scalp | Stratum: Periphery
Number analyzed (Participants) | 15 | 15
ng/mL
  0.5h | 0.2820 (2.2288) | 0.2199 (3.7060)
  1h | 0.3078 (1.9993) | 0.1957 (2.8664)
  1.5h | 0.2176 (2.8671) | 0.3022 (1.7326)
  2h | 0.1497 (3.0551) | 0.2265 (4.3780)
  2.5h | 0.1634 (2.2679) | 0.3389 (1.8265)
  3h | 0.1369 (2.5145) | 0.1972 (2.2296)
  3.5h | 0.2313 (1.5809) | 0.2334 (3.4067)
  4h | 0.2021 (2.7651) | 0.3522 (3.1629)
  5h | 0.2631 (3.2208) | 0.2344 (2.7834)
  6h | 0.3091 (2.9830) | 0.2076 (2.0474)
  8h | 0.4032 (3.1133) | 0.1863 (3.4056)
  10h | 0.7918 (3.4587) | 0.06873 (3.0953)

3. Secondary Outcome: Evaluation of Baseline-adjusted Pharmacokinetic Parameters of ALA.
Description: Parameter: AUC(0-t) (Area Under Curve); area under the baseline-adjusted plasma concentration-time curve from time zero to the last sampling time point at which the concentration was at or above lower limit of quantification; t(last) is defined as the last value >0 after baseline adjustment.
Time Frame: On treatment day (day 0): 0.5, 1, 1.5, 2, 2.5, 3*, 3.5, 4, 5, 6, 8, 10 hours post-dose (*prior to illumination)
Population: as for outcome 1
Measure: Geometric Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Stratum: Face/Scalp | Stratum: Periphery
Number analyzed (Participants) | 16 | 15
h*ng/mL | 110.03 (2.0) | 71.12 (3.5)

4. Secondary Outcome: Evaluation of Baseline-adjusted Pharmacokinetic Parameters of ALA.
Description: Parameter: AUC(0-∞) (Area Under Curve); area under the baseline-adjusted plasma concentration-time data extrapolated to infinity
Time Frame: On treatment day (day 0): 0.5, 1, 1.5, 2, 2.5, 3*, 3.5, 4, 5, 6, 8, 10 hours post-dose (*prior to illumination)
Population: as for outcome 1
Measure: Geometric Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Stratum: Face/Scalp | Stratum: Periphery
Number analyzed (Participants) | 6 | 3
h*ng/mL | 138.41 (2.2) | 138.55 (1.9)

5. Secondary Outcome: Evaluation of Baseline-adjusted Pharmacokinetic Parameters of ALA.
Description: Parameter: %AUC(t-∞) (Area Under Curve); proportion of extrapolated part
Time Frame: On treatment day (day 0): 0.5, 1, 1.5, 2, 2.5, 3*, 3.5, 4, 5, 6, 8, 10 hours post-dose (*prior to illumination)
Population: as for outcome 1
Measure: Geometric Mean (Standard Deviation); unit: percentage of AUC (0-∞)
Arm/Group | Stratum: Face/Scalp | Stratum: Periphery
Number analyzed (Participants) | 9 | 3
percentage of AUC (0-∞) | 8.27 (2.3) | 3.01 (2.6)

6. Secondary Outcome: Evaluation of Baseline-adjusted Pharmacokinetic Parameters of ALA.
Description: Parameter: Cmax (Maximum Plasma Concentration); observed maximum baseline-adjusted plasma concentration
Time Frame: On treatment day (day 0): 0.5, 1, 1.5, 2, 2.5, 3*, 3.5, 4, 5, 6, 8, 10 hours post-dose (*prior to illumination)
Population: as for outcome 1
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | Stratum: Face/Scalp | Stratum: Periphery
Number analyzed (Participants) | 16 | 15
ng/mL | 27.93 (1.9) | 27.68 (4.1)

7. Secondary Outcome: Evaluation of Baseline-adjusted Pharmacokinetic Parameters of ALA.
Description: Parameter: Tmax (time to reach Cmax)
Time Frame: On treatment day (day 0): 0.5, 1, 1.5, 2, 2.5, 3*, 3.5, 4, 5, 6, 8, 10 hours post-dose (*prior to illumination)
Population: as for outcome 1
Measure: Median (Full Range); unit: h
Arm/Group | Stratum: Face/Scalp | Stratum: Periphery
Number analyzed (Participants) | 16 | 15
h | 3.0 [1.55 to 3.5] | 3.42 [0.47 to 6.0]

8. Secondary Outcome: Evaluation of Baseline-adjusted Pharmacokinetic Parameters of ALA.
Description: Parameter: λz (Elimination Rate Constant); λz denotes the terminal rate constant estimated by linear regression analysis from a range of concentrations in the terminal phase estimated for each treatment and subject by log-linear regression from the linear portion of the logarithmic transformed concentration-time plot. The algorithm will start with the last 3 points with quantifiable concentrations and increases the number of involved points by 1 until the time point after Cmax restricted on time points after removing of the BF-200 ALA gel (all PK samples after the gel is wiped off [after 3h±10 min); λz was only determined in subjects in which the log-linear terminal phase could clearly be defined. Resulting unreliable parameters were flagged accordingly and not used in descriptive statistics. If any pharmacokinetic parameter should have been classified as unreliable, all calculations that use this parameter were considered missing.
Time Frame: On treatment day (day 0): 0.5, 1, 1.5, 2, 2.5, 3*, 3.5, 4, 5, 6, 8, 10 hours post-dose (*prior to illumination)
Population: as for outcome 1
Measure: Geometric Mean (Standard Deviation); unit: 1/h
Arm/Group | Stratum: Face/Scalp | Stratum: Periphery
Number analyzed (Participants) | 9 | 3
1/h | 0.24 (1.9) | 0.36 (1.9)

9. Secondary Outcome: Evaluation of Baseline-adjusted Pharmacokinetic Parameters of ALA.
Description: Parameter: t1/2 (apparent terminal half-life); calculated by ln2/λz; t1/2 was only determined in subjects in which the log-linear terminal phase could clearly be defined. Resulting unreliable parameters were flagged accordingly and not used in descriptive statistics. If any pharmacokinetic parameter should have been classified as unreliable, all calculations that use this parameter were considered missing.
Time Frame: On treatment day (day 0): 0.5, 1, 1.5, 2, 2.5, 3*, 3.5, 4, 5, 6, 8, 10 hours post-dose (*prior to illumination)
Population: as for outcome 1
Measure: Geometric Mean (Standard Deviation); unit: h
Arm/Group | Stratum: Face/Scalp | Stratum: Periphery
Number analyzed (Participants) | 9 | 3
h | 2.86 (1.9) | 1.93 (1.9)

10. Secondary Outcome: Evaluation of Baseline-adjusted Pharmacokinetic Parameters of PpIX.
Description: as for outcome 3
Time Frame: On treatment day (day 0): 0.5, 1, 1.5, 2, 2.5, 3*, 3.5, 4, 5, 6, 8, 10 hours post-dose (*prior to illumination)
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Stratum: Face/Scalp | Stratum: Periphery
Number analyzed (Participants) | 13 | 9
h*ng/mL | 0.88 (4.6) | 0.68 (4.4)

11. Secondary Outcome: Evaluation of Baseline-adjusted Pharmacokinetic Parameters of PpIX.
Description: as for outcome 4
Time Frame: On treatment day (day 0): 0.5, 1, 1.5, 2, 2.5, 3*, 3.5, 4, 5, 6, 8, 10 hours post-dose (*prior to illumination)
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Stratum: Face/Scalp | Stratum: Periphery
Number analyzed (Participants) | 0 | 1
h*ng/mL |  | 0.77 (0)

12. Secondary Outcome: Evaluation of Baseline-adjusted Pharmacokinetic Parameters of PpIX.
Description: Parameter: %AUC(t-∞) (Area Under Curve); proportion of extrapolated part
Time Frame: On treatment day (day 0): 0.5, 1, 1.5, 2, 2.5, 3*, 3.5, 4, 5, 6, 8, 10 hours post-dose (*prior to illumination)
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: percentage of AUC (0-∞)
Arm/Group | Stratum: Face/Scalp | Stratum: Periphery
Number analyzed (Participants) | 0 | 1
percentage of AUC (0-∞) |  | 7.33 (0)

13. Secondary Outcome: Evaluation of Baseline-adjusted Pharmacokinetic Parameters of PpIX.
Description: Parameter: Cmax (Maximum Plasma Concentration); observed maximum baseline-adjusted plasma concentration
Time Frame: On treatment day (day 0): 0.5, 1, 1.5, 2, 2.5, 3*, 3.5, 4, 5, 6, 8, 10 hours post-dose (*prior to illumination)
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | Stratum: Face/Scalp | Stratum: Periphery
Number analyzed (Participants) | 13 | 9
ng/mL | 0.48 (2.2) | 0.34 (2.2)

14. Secondary Outcome: Evaluation of Baseline-adjusted Pharmacokinetic Parameters of PpIX.
Description: Parameter: Tmax (time to reach Cmax)
Time Frame: On treatment day (day 0): 0.5, 1, 1.5, 2, 2.5, 3*, 3.5, 4, 5, 6, 8, 10 hours post-dose (*prior to illumination)
Population: as for outcome 2
Measure: Median (Full Range); unit: h
Arm/Group | Stratum: Face/Scalp | Stratum: Periphery
Number analyzed (Participants) | 13 | 9
h | 4.0 [1.0 to 9.88] | 3.52 [0.47 to 8.0]

15. Secondary Outcome: Evaluation of Baseline-adjusted Pharmacokinetic Parameters of PpIX.
Description: as for outcome 8
Time Frame: On treatment day (day 0): 0.5, 1, 1.5, 2, 2.5, 3*, 3.5, 4, 5, 6, 8, 10 hours post-dose (*prior to illumination)
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: 1/h
Arm/Group | Stratum: Face/Scalp | Stratum: Periphery
Number analyzed (Participants) | 0 | 1
1/h |  | 0.35 (0)

16. Secondary Outcome: Evaluation of Baseline-adjusted Pharmacokinetic Parameters of PpIX.
Description: as for outcome 9
Time Frame: On treatment day (day 0): 0.5, 1, 1.5, 2, 2.5, 3*, 3.5, 4, 5, 6, 8, 10 hours post-dose (*prior to illumination)
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: h
Arm/Group | Stratum: Face/Scalp | Stratum: Periphery
Number analyzed (Participants) | 0 | 1
h |  | 1.95 (0)

17. Secondary Outcome: Assessment of the Frequency and Severity of All Treatment-emergent Adverse Events (TEAEs), Including Serious Adverse Events (SAEs) in Response to PDT With BF-200 ALA Under Maximal Use Conditions.
Description: Frequency of treatment-emergent adverse events (TEAEs),including serious adverse events (SAEs).
Time Frame: On treatment day until end of study approximately 4 weeks after treatment day (day 0)
Population: Safety analysis set (SAF): includes all subjects who underwent at least one of the following treatment procedures: preparation of the treatment field(s), application of BF-200 ALA, or illumination. If the conduct of any treatment procedures was not certain, the subject was to be included in the SAF.
Measure: Count of Participants; unit: Participants
Arm/Group | Stratum: Face/Scalp | Stratum: Periphery
Number analyzed (Participants) | 16 | 16
Participants
  Application site erythema | 16 | 16
  Application site exfoliation | 10 | 3
  Application site hyperaesthesia | 2 | 2
  Application site induration | 2 | 2
  Application site oedema | 16 | 9
  Application site pain | 16 | 16
  Application site paraesthesia | 4 | 1
  Application site pruritus | 4 | 6
  Application site scab | 5 | 6
  Application site vesicles | 1 | 2
  Application site warmth | 4 | 1

18. Secondary Outcome: Assessment of Pain Intensity at the Application Site in Response to PDT With BF-200 ALA Under Maximal Use Conditions Using an 11-point Numeric Rating Scale (NRS-11), Where a Score of 0 Means "no Pain" and a Score of 10 Means "Worst Imaginable Pain".
Description: Assessment of pain at the application site using an 11-point Numeric Rating Scale (NRS-11) ranging from 0 (no pain) to 10 (worst imaginable pain)
Time Frame: On treatment day until end of study approximately 4 weeks after treatment day (day 0)
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stratum: Face/Scalp | Stratum: Periphery
Number analyzed (Participants) | 16 | 16
score on a scale | 8.1 (2.0) | 6.0 (2.1)

19. Secondary Outcome: Assessment of Frequency and Severity of Application Site Discomfort in Response to PDT With BF-200 ALA Under Maximal Use Conditions.
Description: Application site reactions: discomfort (burning, pain, itching, stinging, warmth, others)
Time Frame: On treatment day until end of study approximately 4 weeks after treatment day (day 0)
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Stratum: Face/Scalp | Stratum: Periphery
Number analyzed (Participants) | 16 | 16
Participants
  Burning | 14 | 9
  Itching | 4 | 6
  Other | 8 | 1
  Pain | 15 | 7
  Pain during PDT | 16 | 16
  Stinging | 7 | 3
  Warmth | 4 | 1

20. Secondary Outcome: Assessment of Frequency and Severity of Application Site Skin Reactions in Response to PDT With BF-200 ALA Under Maximal Use Conditions.
Description: Application site reactions: skin reactions (erythema, edema, induration, vesicles, erosion, ulceration, scaling/flaking, scabbing/crusting, discharge/exudate, others); maximum severity of AE: mild, moderate, or severe
Time Frame: On treatment day until end of study approximately 4 weeks after treatment day (day 0)
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Stratum: Face/Scalp | Stratum: Periphery
Number analyzed (Participants) | 16 | 16
Participants
  Discharge/exudate | 1 | 0
  Oedema | 16 | 9
  Erythema | 16 | 16
  Induration | 2 | 2
  Other | 12 | 4
  Scabbing/crusting | 5 | 6
  Scaling/flaking | 2 | 3

ADVERSE EVENTS:
Time Frame: On treatment day until end of study approximately 4 weeks after treatment day (07 October 2020, study completion date).
Description: TEAEs (treatment emergent adverse events) are defined as all AEs or SAEs that occurred after lesion preparation at Visit 2, which was at maximum one hour before IMP application (i.e. AE onset date/time ≥ date/time of IMP application (Visit 2) - 1 h).
Arm/Group | Stratum: Face/Scalp | Stratum: Periphery
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 16/16 | 16/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stratum: Face/Scalp (N=16) | Stratum: Periphery (N=16)
Application site erythema (General disorders) | 16 (18) | 16 (19)
Application site exfoliation (General disorders) | 10 (13) | 3 (4)
Application site hyperaesthesia (General disorders) | 2 (3) | 1 (2)
Application site induration (General disorders) | 2 (3) | 2 (2)
Application site oedema (General disorders) | 16 (18) | 9 (10)
Application site pain (General disorders) | 16 (63) | 16 (44)
Application site paraesthesia (General disorders) | 4 (5) | 1 (2)
Application site pruritus (General disorders) | 4 (4) | 6 (7)
Application site scab (General disorders) | 5 (6) | 6 (6)
Application site vesicles (General disorders) | 1 (1) | 2 (4)
Application site warmth (General disorders) | 4 (5) | 1 (1)
Application site discharge (General disorders) | 1 (1) | 0 (0)
Application site discolouration (General disorders) | 1 (1) | 1 (1)
Application site erosion (General disorders) | 1 (1) | 1 (1)
Application site fissure (General disorders) | 1 (2) | 1 (2)
Application site haemorrhage (General disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Seasonal allergy (Immune system disorders) | 1 (1) | 0 (0)
Application site pustules (Infections and infestations) | 1 (2) | 0 (0)
Bacteriuria (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0)
Pyuria (Infections and infestations) | 1 (1) | 0 (0)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Sinus headache (Nervous system disorders) | 1 (1) | 0 (0)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
It is understood that no results or data shall be independently published by the Principal Investigator, the Institution, or its other Representatives prior to Sponsor's approval. The Principal Investigator may publish the results of his or her investigative findings under the Study to the extent they are included in the individual Study publication or as part of a comprehensive publication.

DOCUMENTS (2):
  • Study Protocol (2020-01-17): https://cdn.clinicaltrials.gov/large-docs/59/NCT04319159/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-30): https://cdn.clinicaltrials.gov/large-docs/59/NCT04319159/SAP_001.pdf